CLINICAL TRIAL: NCT05752890
Title: Developing a Novel Biomarker for Response and Prognosis of HBV-related Hepatocellular Carcinoma Treated With Radiotherapy: Personalized Cell-free Virus-host Chimera DNA
Brief Title: A Novel Biomarker for Response and Prognosis of HBV-related Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202212021RINB
Record Dates: First submitted 2023-01-30; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma; Hepatitis b Virus; Radiotherapy; Biomarker
Keywords: Hepatocellular Carcinoma; Hepatitis b Virus; Radiotherapy; Chimera DNA; Biomarker
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — We plan to identify HBV integrations by Capture NGS and quantify the specific vh-DNA by ddPCR as personalized biomarkers from the same-patient serum samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will first use our previously collected serum samples and surgical/biopsied tissues from HBV-related HCC patients undergoing radiotherapy. The consistency of junctional clones by Capture NGS needs to be tested between both pre- and post-RT serums, and serial changes in copy numbers of vh-DNA by ddPCR are quantified in the representative cases. The same junction clones from pre-post-RT serums and surgical tissues will be confirmed and the copy number changes of vh-DNA be correlated with RT response and disease-control status.

The investigators plan to identify HBV integrations by Capture NGS and quantify the specific vh-DNA by ddPCR as personalized biomarkers from the same-patient serum samples. The investigators will further correlate clinical response and recurrence/metastasis with serial changes of vh-DNA copy numbers. The investigators have been prospectively collecting plasma samples from HBV-related HCC patients before/after RT, at 1, 4, 7 months, and at recurrence/metastasis. The investigators plan to confirm the viable role of pre-/post-RT changes of plasma vh-DNA copies of the same junction clone in post-RT response and prognosis. Moreover, The investigators will explore the recurrent/metastatic tumors arising from the original or a de novo one by identifying their clonality with HBV integration patterns. The true value of this novel HBV chimera vh-DNA will be revealed. The results will also support the consolidative use of personalized vh-DNA for earlier evaluating treatment response after RT, for post-RT disease monitoring, and for differentiating clonality at recurrence to design future clinical trial on combinational treatment.

DETAILED DESCRIPTION:
Residual tumors and early recurrence/metastasis after radiotherapy (RT) compromise the patient survival with hepatocellular carcinoma (HCC). Timely detecting residual/recurrence/metastasis and the clonality is required to implement salvage therapies properly. The major unmet needs of radiotherapy to HCC are the difficulties in early evaluating response by images and timely detection of intrahepatic recurrence and extrahepatic metastasis. Thus, an accurate and personalized biomarker for response prediction and disease monitoring is demanded. Cell-free tumor-specific DNA (ctDNA) has garnered attention as a promising biomarker in cancer patients. However, in HCC, the detection rate is low (9-21.2%), mainly due to the limited prevalence of traditional somatic mutations and the difficult separation of ctDNA fragments from normal cells. The investigators aim to develop a novel ctDNA, the virus-host chimera DNA (vh-DNA), as a biomarker for hepatitis B virus (HBV)-related HCC patients undergoing RT. HBV vh-DNA presents in ~90% of HBV-related HCC patients and can be differentiated from DNA released from the normal cells through enrichment by capturing with HBV probes. vh-DNA might be advantageous to the traditional somatic mutation type of ctDNA. The investigators hypothesize that HBV vh-DNA could accurately diagnose residual tumor by 6-12 months earlier than contemporary images and predict early recurrence/metastatsis, thus allows early intervention of salvage therapies.

The investigators will first use our previously collected serum samples and surgical/biopsied tissues from HBV-related HCC patients undergoing radiotherapy. The consistency of junctional clones by Capture NGS needs to be tested between both pre- and post-RT serums, and serial changes in copy numbers of vh-DNA by ddPCR are quantified in the representative cases. The same junction clones from pre-post-RT serums and surgical tissues will be confirmed and the copy number changes of vh-DNA be correlated with RT response and disease-control status.

The investigators plan to identify HBV integrations by Capture NGS and quantify the specific vh-DNA by ddPCR as personalized biomarkers from the same-patient serum samples. The investigators will further correlate clinical response and recurrence/metastasis with serial changes of vh-DNA copy numbers. The investigators have been prospectively collecting plasma samples from HBV-related HCC patients before/after RT, at 1, 4, 7 months, and at recurrence/metastasis. The investigators plan to confirm the viable role of pre-/post-RT changes of plasma vh-DNA copies of the same junction clone in post-RT response and prognosis. Moreover, The investigators will explore the recurrent/metastatic tumors arising from the original or a de novo one by identifying their clonality with HBV integration patterns. The true value of this novel HBV chimera vh-DNA will be revealed. The results will also support the consolidative use of personalized vh-DNA for earlier evaluating treatment response after RT, for post-RT disease monitoring, and for differentiating clonality at recurrence to design future clinical trial on combinational treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with HCC by dynamic image criteria and/or biopsy
2. HBsAg (+)
3. Child-Turcotte-Pugh (CTP) class A-B liver function
4. Radiotherapy to liver tumor as the main treatment

Exclusion Criteria:

1. Child-Turcotte-Pugh (CTP) class C liver functiECOG performance status score >2
2. Has had prior radiotherapy to the proposed treatment field.
3. < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: we have been prospectively collecting plasma samples from HBV-related HCC patients before/after RT, at 1, 4, 7 months, and at recurrence/metastasis.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2031-01-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
To retrospectively analyze the Capture-NGS analysis from HBV-related HCC patients | 2031/01/01
  Capture-NGS analysis and identification of HBV-human junction between pre- and post- RT
To retrospectively analyze the Vh-DNA specific PCR from HBV-related HCC patients | 2031/01/01
  Vh-DNA specific PCR between pre- and post- RT
To retrospectively analyze the serial changes of serum vh-DNA copies of same junction clone from HBV-related HCC patients | 2031/01/01
  Treatment response between pre- and post- RT
To retrospectively analyze the serial changes of survival of same junction clone from HBV-related HCC patients | 2031/01/01
  Survival between pre- and post- RT
To prospectively test the concordance of vh-DNA copies between serum and plasma samples | 2031/01/01
  Calculate the percentage of identical vhDNA sets between the simultaneously collected serum and plasma samples in the same patients
To prospectively analyze the serial changes of plasma vh-DNA copies of same junction clone are associated with treatment response | 2031/01/01
  Treatment response will be determined as the best response in serial image follow-ups up to 6 months after completion of RT. Responses will be classified as completion response, partial response, stable disease, and progressive disease by the definition of mRECIST.
To prospectively analyze the serial changes of plasma vh-DNA copies of same junction clone are associated with overall survival | 2031/01/01
  It will be calculated from the last fraction of radiotherapy until death from any cause of last follow-up.
To distinguish the clonality of recurrent HCC as the original or a de novo one for post-radiotherapy patterns of failure | 2031/01/01
  Detected tumor-specific vh-DNA in the plasma collected at the time of recurrence/metastasis to determine its clonality.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsien Cheng, Principal Investigator — Employee